CLINICAL TRIAL: NCT02760758
Title: A Phase Ia/Ib Study Assessing Single and Multiple Doses of CDI-31244: A Non-Nucleoside Inhibitor in Healthy and Hepatitis C Virus-Infected Subjects
Brief Title: A Study of CDI-31244: A Novel NNI in HV and HCV Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cocrystal Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDI-31244-P1-001
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2016-08

CONDITIONS: Hepatitis C
Keywords: non-nucleoside inhibitor; NNI; HCV; DAA
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Cohort 1A HV (Experimental): CDI-31244 20 mg active or placebo single dose (SD)
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 2A HV (Experimental): CDI-31244 50 mg active or placebo SD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 3A HV (Experimental): CDI-31244 100 mg active or placebo SD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 4A HV (Experimental): CDI-31244 200 mg active or placebo SD; food effect
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 5A HV (Experimental): CDI-31244 400 mg active or placebo SD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 6A HV (Experimental): CDI-31244 200 mg active or placebo multiple dose (MD)
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 7A HV (Experimental): CDI-31244 200 mg active or placebo MD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 8A HV (Experimental): CDI-31244 400 mg active or placebo MD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 1B HCV genotype (GT) 1 (Experimental): CDI-31244 400 mg active or placebo MD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 2B HCV GT 1 (Experimental): CDI-31244 600 mg active or placebo MD
  Interventions: Drug: CDI-31244; Drug: Placebo
- Cohort 3B HCV GT 1 (Experimental): CDI-31244 800 mg active or placebo MD
  Interventions: Drug: CDI-31244; Drug: Placebo

INTERVENTIONS:
Drug: CDI-31244 — NNI
  Other Names: CC-31244
Drug: Placebo — no active ingredients
  Other Names: CDI-31244 Placebo

SUMMARY:
This is a First in Human study of orally administered CDI-31244, a non-nucleoside inhibitor (NNI) in healthy volunteers and HCV infected individuals

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo-controlled, randomized, single ascending oral dose and multiple oral dose design, incorporating fed/fasted comparisons.

The study will include two groups: Group A - single ascending dose (SAD) including a food effect cohort, and multiple dose (MD) in healthy volunteers (HV), and Group B MD in Hepatitis C Virus (HCV) infected individuals divided in two parts.

Five single-dose cohort are planned. For the five single-dose cohorts, a sentinel group of 2 subjects will be dosed at least one day prior to enrolling remaining subjects.

Six multiple-dose cohorts are planned. Three multiple dose cohorts in healthy volunteers and three cohorts in HCV-infected individuals.

The dosing of Group B will be conducted following safety and pharmacokinetic (PK) review of Group A. The dosing of Group B, Part 2 will be conducted only if Part 1 shows acceptable safety and efficacy results.

ELIGIBILITY:
Main Inclusion Criteria:

HV and HCV INFECTED SUBJECTS:

* Male or female aged ≥ 18 to ≤ 65 years;
* Body mass index ≥ 18.5 to ≤ 35.0 kg/m2;
* Body weight ≥ 50 kg;
* Negative screening for alcohol and drugs of abuse;
* Normal results on 12-lead electrocardiogram (ECG);
* For females, negative result on a pregnancy test.

HCV INFECTED SUBJECTS:

* HCV treatment-naïve subjects must have not received prior direct acting agent (DAA) treatment for hepatitis C infection;
* Documented clinical history compatible with chronic hepatitis C;
* HCV Genotype 1 by HCV genotyping performed at Screening;
* Plasma HCV RNA ≥ 5.0 log10 IU/mL at Screening;
* Laboratory evidence of no cirrhosis (negative liver biopsy or fibroscan or FibroTest, F2 or lower) within one year prior to study), if these are not available, do a FibroTest at screening, which must be F2 or lower.

Main Exclusion Criteria:

HV and HCV INFECTED SUBJECTS:

* Females who are pregnant or are lactating;
* Co-infected with hepatitis B virus (HBV, HBsAg positive) and/or human immunodeficiency virus (HIV);
* Abuse of alcohol and/or drugs that could interfere with adherence to study requirements as judged by the investigator;
* Positive screen result for drugs of abuse or alcohol on Day -1. Use of other investigational drugs within 60 days of dosing;
* Subject with intestinal malabsorption;
* Presence of out-of-range cardiac interval on the screening ECG or other clinically significant ECG abnormalities;
* Serum creatinine > upper limit of normal (ULN);
* Any clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.

HEALTHY VOLUNTEERS:

* Positive screen for anti-HCV antibody

HCV INFECTED SUBJECTS:

* Clinical (in the opinion of the investigator) or laboratory evidence of cirrhosis;
* History or signs of decompensated liver disease: ascites, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, or other clinical signs of portal hypertension or hepatic insufficiency;
* History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC;
* Active clinically significant diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (AE) | Day 1 to Day 35
  The safety and the tolerability of single and multiple oral doses of CDI-31244 through number of AEs observed in HV and HCV infected subjects

SECONDARY OUTCOMES:
Measure plasma levels of CDI-31244 after SD | Day 1 to Day 6
  Plasma levels of CDI-31244 in the the single dose HV cohorts
Measure plasma levels of CDI-31244 after SD in fasted and fed conditions | Day 1 to Day 13
  The effect of food on the plasma levels of CDI-31244 in the single dose HV cohorts
Measure plasma levels of CDI-31244 after MD | Day 1 to Day 13
  Plasma levels of CDI-31244 in the multiple dose HV and HCV infected cohorts
Measure HCV viral load through the RNA quantitative test | Day 1 to Day 35
  The clinical efficacy of CDI-31244 in HCV-infected subjects as measured by the maximal change in antiviral activity through changes in the HCV RNA load
Measure HCV mutation through genotyping at baseline and after CDI-31244 dosing | Day 1 to 35
  The possible emergence of hepatitis C virus resistance mutation in HCV infected subjects

CONTACTS AND LOCATIONS:
Overall Officials: Judy Pattassery, Study Director — Cocrystal Pharma, Inc.
Locations (1):
- Algorithme, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No